CLINICAL TRIAL: NCT05269095
Title: Analgesic Effect of Adductor Canal Block Combined With Infiltration of the Interspace Between Popliteal Artery and the Capsule of the Knee (IPACK) Block Versus Genicular Nerves Block in Knee Arthroscopy
Brief Title: Adductor Canal Block Combined With IPACK vs Genicular Nerves Block in Knee Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Muhammad Ahmed Kandil, Resident of Anesthesiology and Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35236/1/22
Record Dates: First submitted 2022-03-04; First posted 2022-03-07 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Arthroscopy; Genicular Nerves Block
MeSH Terms: interventions — Anesthesia, Spinal; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- spinal anesthesia only (Experimental): Patients will receive spinal anesthesia only
  Interventions: Procedure: Spinal anesthesia only
- spinal anesthesia and ultrasound-guided Genicular nerves block (Experimental): Patients will receive spinal anesthesia and ultrasound-guided Genicular nerves block
  Interventions: Biological: Spinal anesthesia and ultrasound-guided Genicular nerves block
- Spinal anesthesia and US guided Adductor canal nerve block plus infiltration of the interspace (Experimental): Patients will receive spinal anesthesia and ultrasound-guided Adductor canal nerve block plus infiltration of the interspace between the popliteal artery and the capsule of the posterior knee (PACK) block.
  Interventions: Biological: Ultrasound-guided Adductor Canal block (ACB) technique with infiltration of the interspace between popliteal artery and the capsule of posterior knee block ('PACK)

INTERVENTIONS:
Procedure: Spinal anesthesia only — Patients will receive spinal anesthesia with 2-3 ml 0.5% (10-15 mg) hyperbaric bupivacaine plus 25 ug fentanyl at the L3/4 interspaces.
  Arms: spinal anesthesia only
Biological: Spinal anesthesia and ultrasound-guided Genicular nerves block — Patients will receive16 ml bupivacaine 0025% will be administered, and4 ml of this solution will be placed at each of the 4 target nerves.
  Arms: spinal anesthesia and ultrasound-guided Genicular nerves block
Biological: Ultrasound-guided Adductor Canal block (ACB) technique with infiltration of the interspace between popliteal artery and the capsule of posterior knee block ('PACK) — Adductor Canal block (ACB) technique will be performed using 16 ml bupivacaine 0025% As regarding the Popliteal artery and the capsule of posterior knee block ('PACK), it will be performed Using 16 ml bupivacaine 0.25%
  Arms: Spinal anesthesia and US guided Adductor canal nerve block plus infiltration of the interspace

SUMMARY:
This prospective randomized controlled study is designed to investigate the postoperative analgesic effect of adductor canal block (ACB) combined with infiltration of the interspace between the popliteal artery and the capsule of posterior knee (IPACK) block compared to genicular nerves block in patients undergoing knee arthroscopy.

DETAILED DESCRIPTION:
Maintaining patient safety, ensuring best patient outcomes, and optimal pain relief post-operatively are of utmost concern for anesthesia providers. Adequate pain relief attenuates stress responses and long-term chronic pain complications while contributing to improved postoperative outcomes.

Knee arthroscopy is a very common procedure and very often is performed as day-case surgery. Ambulatory arthroscopic surgery of the knee is preferred by the majority of properly selected and well-informed patients. It has been reported that a significant number of patients have moderate to severe pain 24 hours after ambulatory surgery in general and knee arthroscopy in particular and pain affects the patient's activity level and satisfaction. Adductor canal block (ACB) is a popular peripheral nerve block that has been shown to decrease the pain significantly and decrease opioid consumption with minimal effect on quadriceps function. It provides analgesia to the peri-articular and intra-articular aspects of the knee joint but doesn't relieve posterior knee pain which is moderate to severe in intensity.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60 years
* Both genders
* American Society of Anaesthesiologists physical status classification I - III
* Patients scheduled for elective unilateral knee arthroscopy under spinal anesthesia

Exclusion Criteria:

* Patient refusal
* Preoperative neurological deficits
* Opioid-dependent (opioid intake more than 3 months)
* Chronic pain conditions
* Significant cardiac and respiratory disease
* Pre-existing major organ dysfunction such as hepatic and renal failure
* Coexisting hematological disorder or deranged coagulation parameters
* Psychiatric illnesses
* Allergy to any of the drugs used in the study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-03-21 (Estimated); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-03-21 (Estimated)

PRIMARY OUTCOMES:
Postoperative 24-hour rescue analgesic consumption | 24 hours postoperative
  Total postoperative 24-hour rescue analgesic consumption will be recorded

SECONDARY OUTCOMES:
Post-operative pain | 24 hours Postoperative
  Post-operative pain will be assessed by the Numeric Rating Scale (NRS) rest and mobilization.
Time taken till 1st rescue analgesic request | 24 hours Postoperative
  The time till administration of first rescue analgesia will be recorded

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study